CLINICAL TRIAL: NCT00289731
Title: Evaluate the Effect of Several Risk Factors That Are Likely to Influence the Immunogenicity of GSK Biologicals' Combined Hepatitis A & B Vaccine, vs Separately Administered Monovalent Hepatitis A and Hepatitis B Vaccines
Brief Title: Effect of Risk Factors Likely to Influence Immuno of Combined Hepatitis A & B Vacc vs Monovalent Hepatitis A & B Vacc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100382; 100383 (Other: GSK); 100384 (Other: GSK); 100385 (Other: GSK)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Hepatitis B; Hepatitis A
Keywords: Combined hepatitis A and hepatitis B vaccine; Hepatitis B; Hepatitis A; Monovalent hepatitis A and hepatitis B vaccines
MeSH Terms: conditions — Hepatitis B; Hepatitis A | interventions — twinrix; Hepatitis A Vaccines

ARMS (3):
- Twinrix Group (Experimental): Healthy and non-healthy male or female subjects, aged 41 years or older, who received combined Twinrix™ (720/20) vaccine, administered intramuscularly in the left deltoid region, according to a 0, 1 and 6 month schedule.
  Interventions: Biological: TWINRIX™
- Engerix-B+Havrix Group (Active Comparator): Healthy and non-healthy male or female subjects, aged 41 years or older, who received separate administrations of Engerix™-B (20 μg) vaccine, administered intramuscularly in the left deltoid region, according to a 0, 1 and 6 month schedule and Havrix™ (1440 EL.U) vaccine, administered intramuscularly in the right deltoid region, according to a 0 and 6 month schedule.
  Interventions: Biological: Engerix™-B; Biological: HAVRIX™
- HB VAX PRO+Vaqta Group (Active Comparator): Healthy and non-healthy male or female subjects, aged 41 years or older, who received separate administrations of HB VAX PRO™ (10 μg) vaccine, administered intramuscularly in the left deltoid region, according to a 0, 1 and 6 month schedule and Vaqta™ (50 IU) vaccine, administered intramuscularly in the right deltoid region, according to a 0 and 6 month schedule.
  Interventions: Biological: HB VAX PRO™; Biological: Vaqta™

INTERVENTIONS:
Biological: TWINRIX™ — Intramuscular injection, 3 doses
  Arms: Twinrix Group
Biological: Engerix™-B — Intramuscular injection, 3 doses
  Arms: Engerix-B+Havrix Group
Biological: HAVRIX™ — Intramuscular injection, 2 doses
  Arms: Engerix-B+Havrix Group
Biological: HB VAX PRO™ — Intramuscular injection, 3 doses
  Arms: HB VAX PRO+Vaqta Group
Biological: Vaqta™ — Intramuscular injection, 2 doses
  Arms: HB VAX PRO+Vaqta Group

SUMMARY:
The focus of this study is to evaluate how risk factors like age, gender, body mass index, smoking, alcohol consumption, etc. can influence immune response when subjects are vaccinated with GSK Biologicals' combined hepatitis A/hepatitis B vaccine or monovalent hepatitis A and B vaccines (from GSK Biologicals' or different manufacturers). The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The study will also evaluate the persistence of hepatitis A and hepatitis B antibodies at months 12, 24 and 36 after the first dose of primary vaccination course.

ELIGIBILITY:
Inclusion criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* Healthy and non-healthy male or female aged 41 years or older at the time of the first vaccination.
* Written informed consent obtained from the subject.
* No serological signs of hepatitis A or B infection at screening.
* If the subject is female, she must be of non-childbearing potential or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* History of any hepatitis A or hepatitis B vaccination or infection, since the primary vaccination study 100382.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment. .
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions during the primary vaccination period.

Min Age: 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2003-11-24 (Actual); Primary Completion 2004-12-21 (Actual); Study Completion 2004-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- GSK Investigational Site, Wilrijk, Belgium
- GSK Investigational Site, Hradec Králové, Czechia
- Germany (7):
  - GSK Investigational Site, Finsterwalde, Brandenburg
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Geringswalde, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Elmshorn, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=2175

REFERENCES:
- [Background] Van der Wielen M, Van Damme P, Chlibek R, Smetana J, von Sonnenburg F. Hepatitis A/B vaccination of adults over 40 years old: comparison of three vaccine regimens and effect of influencing factors. Vaccine. 2006 Jun 29;24(26):5509-15. doi: 10.1016/j.vaccine.2006.04.016. Epub 2006 May 4. PMID 16725234
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 100382 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100382 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100382 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 100382 are summarised with studies 100383, 100384, and 100385 on the GSK Clinical Study Register.
- Available data/document: Clinical Study Report: 100382 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100382 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100382 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 596 subjects (199 in Twinrix Group, 200 in Engerix-B+Havrix Group and 197 in HB VAX PRO+Vaqta Group) were enrolled and vaccinated in the study.
Groups:
- Twinrix Group: Healthy and non-healthy male or female subjects, aged 41 years or older, who received combined Twinrix (720/20) vaccine, administered intramuscularly in the left deltoid region, according to a 0, 1 and 6 month schedule.
- Engerix-B+Havrix Group: Healthy and non-healthy male or female subjects, aged 41 years or older, who received separate administrations of Engerix-B (20 μg) vaccine, administered intramuscularly in the left deltoid region, according to a 0, 1 and 6 month schedule and Havrix (1440 EL.U) vaccine, administered intramuscularly in the right deltoid region, according to a 0 and 6 month schedule.
- HB VAX PRO+Vaqta Group: Healthy and non-healthy male or female subjects, aged 41 years or older, who received separate administrations of HB VAX PRO (10 μg) vaccine, administered intramuscularly in the left deltoid region, according to a 0, 1 and 6 month schedule and Vaqta (50 IU) vaccine, administered intramuscularly in the right deltoid region, according to a 0 and 6 month schedule.
Period: Overall Study
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Started | 199 | 200 | 197
Completed | 197 | 198 | 195
Not Completed | 2 | 2 | 2
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group | Total
Number analyzed (Participants) | 199 | 200 | 197 | 596
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (9.24) | 55.3 (9.91) | 55.0 (9.64) | 55.17 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 100 | 101 | 298
  Male | 102 | 100 | 96 | 298
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 199 | 200 | 196 | 595
  Black | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations for Anti-hepatitis A Virus (Anti-HAV) and Anti-hepatitis B Surface (Anti-HBs) Antigens
Description: Anti-HAV and anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL). The reference seropositivity cut-off values for anti-HAV and anti-HBs antibodies were equal to or above (≥) 15 mIU/mL and ≥ 3.3 mIU/mL, respectively.
Time Frame: At Month 7 after Twinrix vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all subjects who met all eligibility criteria and for whom data concerning immunogenicity endpoint measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group
Number analyzed (Participants) | 181
mIU/mL
  Anti-HAV | 2746.5 [2256.3 to 3343.2]
  Anti-HBs | 1153.9 [829.8 to 1604.7]

2. Primary Outcome: Number of Subjects With Anti-HAV and Anti-HBs Antibody Concentrations Above the Cut-off Value
Description: Seropositivity for anti-HAV antibodies was defined as anti-HAV antibody concentration ≥ 15mIU/mL; seropositivity for anti-HBs antibodies was defined as anti-HBs antibody concentration ≥ 3.3 mIU/mL.
Time Frame: At Month 7
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all subjects who met all eligibility criteria and for whom data concerning immunogenicity endpoint measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Anti-HAV | 176 | 180 | 174
  Anti-HBs | 168 | 152 | 137
Statistical Analysis 1: Comparison: Twinrix Group vs Engerix-B+Havrix Group; Difference in seropositivity rates against hepatitis A virus (HAV) antigen: To demonstrate that the immunogenicity of Twinrix vaccine (Twinrix Group) administered at Months 0, 1 and 6 was non-inferior to that of separately administered monovalent vaccines Engerix-B at Months 0, 1 and 6 and Havrix at Months 0 and 6 (Engerix-B+Havrix Group), in terms of anti-HAV seropositivity rates, at Month 7; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two treatment groups (Twinrix Group minus Engerix-B+Havrix Group), in terms of seropositivity rates for anti-HAV antibody, being - 10%; Difference in seropositivity rate = -1.66, 95% CI 2-sided [-5.34 to 1.48]
Statistical Analysis 2: Comparison: Twinrix Group vs HB VAX PRO+Vaqta Group; Difference in seropositivity rates against hepatitis A virus (HAV) antigen: To demonstrate that the immunogenicity of Twinrix vaccine (Twinrix Group) administered at Months 0, 1 and 6 was non-inferior to that of separately administered monovalent vaccines HB VAX PRO at Months 0, 1 and 6 and Vaqta at Months 0 and 6 (HB VAX PRO+Vaqta Group), in terms of anti-HAV seropositivity rates, at Month 7; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two treatment groups (Twinrix Group minus HB VAX PRO+Vaqta Group), in terms of seropositivity rates for anti-HAV antibody, being - 10%; Difference in seropositivity rate = -1.63, 95% CI 2-sided [-5.31 to 1.60]

3. Primary Outcome: Number of Seroprotected Subjects Against Hepatitis B Surface (HBs) Antigen
Description: A seroprotected subject was defined as a vaccinated subject with a serum anti-HBs antibody concentration equal to or above (≥) 10 mIU/mL.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants | 166 | 145 | 125
Statistical Analysis 1: Comparison: Twinrix Group vs Engerix-B+Havrix Group; Difference in seroprotection rates against hepatitis B surface (HBs) antigen: To demonstrate that the immunogenicity of Twinrix vaccine (Twinrix Group) administered at Months 0, 1 and 6 was non-inferior to that of separately administered monovalent vaccines Engerix-B at Months 0, 1 and 6 and Havrix at Months 0 and 6 (Engerix-B+Havrix Group), in terms of anti-HBs seroprotection rates, at Month 7; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two treatment groups (Twinrix Group minus Engerix-B+Havrix Group), in terms of seroprotection rates for anti-HBs antibody, being - 10%; Difference in seroprotection rate = 12.04, 95% CI 2-sided [4.97 to 19.35]
Statistical Analysis 2: Comparison: Twinrix Group vs HB VAX PRO+Vaqta Group; Difference in seropositivity rates against hepatitis B surface (HBs) antigen: To demonstrate that the immunogenicity of Twinrix vaccine (Twinrix Group) administered at Months 0, 1 and 6 was non-inferior to that of separately administered monovalent vaccines HB VAX PRO at Months 0, 1 and 6 and Vaqta at Months 0 and 6 (HB VAX PRO+Vaqta Group), in terms of anti-HBs seroprotection rates, at Month 7; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two treatment groups (Twinrix Group minus HB VAX PRO+Vaqta Group), in terms of seroprotection rates for anti-HBs antibody, being - 15%; Difference in seroprotection rates = 20.69, 95% CI 2-sided [12.92 to 28.62]

4. Secondary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations
Description: as for outcome 1
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 168 | 165
mIU/mL
  Anti-HAV | 1394.3 [1159.8 to 1676.1] | 3707.2 [3081.4 to 4460.2]
  Anti-HBs | 491.2 [342.3 to 704.9] | 179.1 [128.5 to 249.7]

5. Secondary Outcome: Number of Subjects With Anti-HAV and Anti-HBs Antibody Concentrations Above the Cut-off Value, by Gender
Description: Seropositivity for anti-HAV antibodies was defined as anti-HAV antibody concentration equal to or above (≥) 15 mIU/mL and anti-HBs seropositivity was defined as anti-HBs antibody concentrations ≥ 3.3 mIU/mL. The seropositivity rates were stratified by gender (females and males).
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Anti-HAV, Females: number analyzed (Participants) | 88 | 89 | 90
  Anti-HAV, Females | 86 | 88 | 89
  Anti-HAV, Males: number analyzed (Participants) | 93 | 93 | 86
  Anti-HAV, Males | 90 | 92 | 85
  Anti-HBs, Females: number analyzed (Participants) | 88 | 89 | 90
  Anti-HBs, Females | 82 | 77 | 78
  Anti-HBs, Males: number analyzed (Participants) | 93 | 93 | 86
  Anti-HBs, Males | 86 | 75 | 59

6. Secondary Outcome: Number of Subjects With Anti-HAV and Anti-HBs Antibody Concentrations Above the Cut-off Value, by Age
Description: Seropositivity for anti-HAV antibodies was defined as anti-HAV antibody concentration equal to or above (≥) 15 mIU/mL and anti-HBs seropositivity was defined as anti-HBs antibody concentrations ≥ 3.3 mIU/mL. The seropositivity rates were stratified by age as follows: ≤ 50 years of age (YOA), 51-60 YOA and ≥ 61 YOA.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Anti-HAV, ≤ 50 YOA: number analyzed (Participants) | 59 | 59 | 59
  Anti-HAV, ≤ 50 YOA | 58 | 59 | 59
  Anti-HAV, 51-60 YOA: number analyzed (Participants) | 65 | 64 | 57
  Anti-HAV, 51-60 YOA | 63 | 63 | 57
  Anti-HAV, ≥ 61 YOA: number analyzed (Participants) | 57 | 59 | 60
  Anti-HAV, ≥ 61 YOA | 55 | 58 | 58
  Anti-HBs, ≤ 50 YOA: number analyzed (Participants) | 59 | 59 | 59
  Anti-HBs, ≤ 50 YOA | 57 | 50 | 54
  Anti-HBs, 51-60 YOA: number analyzed (Participants) | 65 | 64 | 57
  Anti-HBs, 51-60 YOA | 63 | 58 | 46
  Anti-HBs, ≥ 61 YOA: number analyzed (Participants) | 57 | 59 | 60
  Anti-HBs, ≥ 61 YOA | 48 | 44 | 37

7. Secondary Outcome: Number of Subjects With Anti-HAV and Anti-HBs Antibody Concentrations Above the Cut-off Value, by Body Mass Index (BMI)
Description: Seropositivity for anti-HAV antibodies was defined as anti-HAV antibody concentration equal to or above (≥) 15 mIU/mL and anti-HBs seropositivity was defined as anti-HBs antibody concentrations ≥ 3.3 mIU/mL. The seropositivity rates were stratified by BMI as follows: healthy, overweight and obese.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Anti-HAV, Healthy: number analyzed (Participants) | 57 | 61 | 58
  Anti-HAV, Healthy | 57 | 61 | 58
  Anti-HAV, Overweight: number analyzed (Participants) | 66 | 63 | 58
  Anti-HAV, Overweight | 66 | 63 | 58
  Anti-HAV, Obese: number analyzed (Participants) | 58 | 58 | 60
  Anti-HAV, Obese | 53 | 56 | 58
  Anti-HBs, Healthy: number analyzed (Participants) | 57 | 61 | 58
  Anti-HBs, Healthy | 53 | 54 | 48
  Anti-HBs, Overweight: number analyzed (Participants) | 66 | 63 | 58
  Anti-HBs, Overweight | 62 | 53 | 44
  Anti-HBs, Obese: number analyzed (Participants) | 58 | 58 | 60
  Anti-HBs, Obese | 53 | 45 | 45

8. Secondary Outcome: Number of Subjects With Anti-HAV and Anti-HBs Antibody Concentrations Above the Cut-off Value, by Smoking Status
Description: Seropositivity for anti-HAV antibodies was defined as anti-HAV antibody concentration equal to or above (≥) 15 mIU/mL and anti-HBs seropositivity was defined as anti-HBs antibody concentrations ≥ 3.3 mIU/mL. The seropositivity rates were stratified by smoking status (smokers and non-smokers).
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Anti-HAV, Smokers: number analyzed (Participants) | 51 | 51 | 32
  Anti-HAV, Smokers | 50 | 51 | 32
  Anti-HAV, Non-smokers: number analyzed (Participants) | 130 | 131 | 144
  Anti-HAV, Non-smokers | 126 | 129 | 142
  Anti-HBs, Smokers: number analyzed (Participants) | 51 | 51 | 32
  Anti-HBs, Smokers | 47 | 44 | 23
  Anti-HBs, Non-smokers: number analyzed (Participants) | 130 | 131 | 144
  Anti-HBs, Non-smokers | 121 | 108 | 114

9. Secondary Outcome: Number of Subjects With Anti-HAV and Anti-HBs Antibody Concentrations Above the Cut-off Value, by Alcohol Consumption
Description: Seropositivity for anti-HAV antibodies was defined as anti-HAV antibody concentration equal to or above (≥) 15 mIU/mL and anti-HBs seropositivity was defined as anti-HBs antibody concentrations ≥ 3.3 mIU/mL. The seropositivity rates were stratified by alcohol consumption as follows: None or Mild, Moderate and Heavy.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Anti-HAV, None or Mild: number analyzed (Participants) | 112 | 106 | 102
  Anti-HAV, None or Mild | 108 | 105 | 100
  Anti-HAV, Moderate: number analyzed (Participants) | 56 | 68 | 62
  Anti-HAV, Moderate | 55 | 67 | 62
  Anti-HAV, Heavy: number analyzed (Participants) | 13 | 8 | 12
  Anti-HAV, Heavy | 13 | 8 | 12
  Anti-HBs, None or Mild: number analyzed (Participants) | 112 | 106 | 102
  Anti-HBs, None or Mild | 105 | 89 | 80
  Anti-HBs, Moderate: number analyzed (Participants) | 56 | 68 | 62
  Anti-HBs, Moderate | 52 | 57 | 47
  Anti-HBs, Heavy: number analyzed (Participants) | 13 | 8 | 12
  Anti-HBs, Heavy | 11 | 6 | 10

10. Secondary Outcome: Number of Subjects With Anti-HAV and Anti-HBs Antibody Concentrations Above the Cut-off Value, by Concomitant Medication
Description: Seropositivity for anti-HAV antibodies was defined as anti-HAV antibody concentration equal to or above (≥) 15 mIU/mL and anti-HBs seropositivity was defined as anti-HBs antibody concentrations ≥ 3.3 mIU/mL. The seropositivity rates were stratified by concomitant medication (concomitant medication and no concomitant medication).
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Anti-HAV, Concomitant medication: number analyzed (Participants) | 165 | 169 | 162
  Anti-HAV, Concomitant medication | 160 | 167 | 160
  Anti-HAV, No concomitant medication: number analyzed (Participants) | 16 | 13 | 14
  Anti-HAV, No concomitant medication | 16 | 13 | 14
  Anti-HBs, Concomitant medication: number analyzed (Participants) | 165 | 169 | 162
  Anti-HBs, Concomitant medication | 153 | 141 | 127
  Anti-HBs, No concomitant medication: number analyzed (Participants) | 16 | 13 | 14
  Anti-HBs, No concomitant medication | 15 | 11 | 10

11. Secondary Outcome: Number of Subjects With Anti-HAV and Anti-HBs Antibody Concentrations Above the Cut-off Value, by Medical Condition
Description: Seropositivity for anti-HAV antibodies was defined as anti-HAV antibody concentration equal to or above (≥) 15 mIU/mL and anti-HBs seropositivity was defined as anti-HBs antibody concentrations ≥ 3.3 mIU/mL. The seropositivity rates were stratified by medical condition as follows: no medical condition, past medical condition and current medical condition.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Anti-HAV,No Medical condition: number analyzed (Participants) | 24 | 20 | 20
  Anti-HAV,No Medical condition | 24 | 20 | 20
  Anti-HAV,Past Medical condition: number analyzed (Participants) | 13 | 22 | 15
  Anti-HAV,Past Medical condition | 13 | 22 | 15
  Anti-HAV,Current Medical condition: number analyzed (Participants) | 144 | 140 | 141
  Anti-HAV,Current Medical condition | 139 | 138 | 139
  Anti-HBs,No Medical condition: number analyzed (Participants) | 24 | 20 | 20
  Anti-HBs,No Medical condition | 23 | 19 | 15
  Anti-HBs,Past Medical condition: number analyzed (Participants) | 13 | 22 | 15
  Anti-HBs,Past Medical condition | 13 | 18 | 12
  Anti-HBs,Current Medical condition: number analyzed (Participants) | 144 | 140 | 141
  Anti-HBs,Current Medical condition | 132 | 115 | 110

12. Secondary Outcome: Number of Seroprotected Subjects Against HBs Antigen, by Gender
Description: A seroprotected subject was defined as a vaccinated subject with a serum anti-HBs antibody concentration equal to or above (≥) 10 mIU/mL. The seroprotection rates were stratified by gender (females and males).
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Females: number analyzed (Participants) | 88 | 89 | 90
  Females | 82 | 73 | 75
  Males: number analyzed (Participants) | 93 | 93 | 86
  Males | 84 | 72 | 50

13. Secondary Outcome: Number of Seroprotected Subjects Against HBs Antigen, by Age
Description: A seroprotected subject was defined as a vaccinated subject with a serum anti-HBs antibody concentration equal to or above (≥) 10 mIU/mL. The seroprotection rates were stratified by age as follows: ≤ 50 years of age (YOA), 51-60 YOA and ≥ 61 YOA.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  ≤ 50 YOA: number analyzed (Participants) | 59 | 59 | 59
  ≤ 50 YOA | 57 | 48 | 52
  51-60 YOA: number analyzed (Participants) | 65 | 64 | 59
  51-60 YOA | 63 | 55 | 43
  ≥ 61 YOA: number analyzed (Participants) | 57 | 59 | 60
  ≥ 61 YOA | 46 | 42 | 30

14. Secondary Outcome: Number of Seroprotected Subjects Against HBs Antigen, by BMI
Description: A seroprotected subject was defined as a vaccinated subject with a serum anti-HBs antibody concentration equal to or above (≥) 10 mIU/mL. The seroprotection rates were stratified by BMI as follows: healthy, overweight and obese.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Healthy: number analyzed (Participants) | 57 | 61 | 58
  Healthy | 52 | 51 | 46
  Overweight: number analyzed (Participants) | 66 | 63 | 58
  Overweight | 62 | 51 | 40
  Obese: number analyzed (Participants) | 58 | 58 | 60
  Obese | 52 | 43 | 39

15. Secondary Outcome: Number of Seroprotected Subjects Against HBs Antigen, by Smoking Status
Description: A seroprotected subject was defined as a vaccinated subject with a serum anti-HBs antibody concentration equal to or above (≥) 10 mIU/mL. The seroprotection rates were stratified by smoking status (smokers and non-smokers).
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Smokers: number analyzed (Participants) | 51 | 51 | 32
  Smokers | 47 | 42 | 22
  Non-smokers: number analyzed (Participants) | 130 | 131 | 144
  Non-smokers | 119 | 103 | 103

16. Secondary Outcome: Number of Seroprotected Subjects Against HBs Antigen, by Alcohol Consumption
Description: A seroprotected subject was defined as a vaccinated subject with a serum anti-HBs antibody concentration equal to or above (≥) 10 mIU/mL. The seroprotection rates were stratified by alcohol consumption as follows: none or mild, moderate and heavy.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  None or Mild: number analyzed (Participants) | 112 | 106 | 102
  None or Mild | 105 | 87 | 76
  Moderate: number analyzed (Participants) | 56 | 68 | 62
  Moderate | 50 | 52 | 41
  Heavy: number analyzed (Participants) | 13 | 8 | 12
  Heavy | 11 | 6 | 8

17. Secondary Outcome: Number of Seroprotected Subjects Against HBs Antigen, by Concomitant Medication
Description: A seroprotected subject was defined as a vaccinated subject with a serum anti-HBs antibody concentration equal to or above (≥) 10 mIU/mL. The seroprotection rates were stratified by concomitant medication (concomitant medication and no concomitant medication).
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  Concomitant medication: number analyzed (Participants) | 165 | 169 | 162
  Concomitant medication | 151 | 135 | 117
  No concomitant medication: number analyzed (Participants) | 16 | 13 | 14
  No concomitant medication | 15 | 10 | 8

18. Secondary Outcome: Number of Seroprotected Subjects Against HBs Antigen, by Medical Condition
Description: A seroprotected subject was defined as a vaccinated subject with a serum anti-HBs antibody concentration equal to or above (≥) 10 mIU/mL. The seroprotection rates were stratified by medical condition as follows: no medical condition, past medical condition and current medical condition.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
Participants
  No medical condition: number analyzed (Participants) | 24 | 20 | 20
  No medical condition | 23 | 18 | 13
  Past medical condition: number analyzed (Participants) | 13 | 22 | 15
  Past medical condition | 13 | 18 | 12
  Current medical condition: number analyzed (Participants) | 144 | 140 | 141
  Current medical condition | 130 | 109 | 100

19. Secondary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations, by Gender
Description: Anti-HAV and anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL). The reference seropositivity cut-off values for anti-HAV and anti-HBs antibodies were equal to or above (≥) 15 mIU/mL and ≥ 3.3 mIU/mL, respectively. The antibody concentrations were stratified by gender (females and males).
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
mIU/mL
  Anti-HAV, Females: number analyzed (Participants) | 88 | 89 | 90
  Anti-HAV, Females | 2968.1 [2176.3 to 4047.9] | 2089.2 [1618.6 to 2696.6] | 5307.0 [4224.5 to 6666.7]
  Anti-HAV, Males: number analyzed (Participants) | 93 | 93 | 86
  Anti-HAV, Males | 2550.3 [1986.6 to 3273.8] | 947.0 [742.2 to 1208.4] | 2546.4 [1932.2 to 3355.8]
  Anti-HBs, Females: number analyzed (Participants) | 88 | 89 | 90
  Anti-HBs, Females | 1957.5 [1295.2 to 2958.4] | 474.2 [274.8 to 818.3] | 273.8 [182.0 to 411.7]
  Anti-HBs, Males: number analyzed (Participants) | 93 | 93 | 86
  Anti-HBs, Males | 697.1 [425.2 to 1142.9] | 509.4 [314.0 to 826.5] | 102.2 [60.1 to 173.8]

20. Secondary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations, by Age
Description: Anti-HAV and anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL). The reference seropositivity cut-off values for anti-HAV and anti-HBs antibodies were equal to or above (≥) 15 mIU/mL and ≥ 3.3 mIU/mL, respectively. The antibody concentrations were stratified by age as follows: ≤ 50 years of age (YOA), 51-60 YOA and ≥ 61 YOA.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
mIU/mL
  Anti-HAV, ≤ 50 YOA: number analyzed (Participants) | 59 | 59 | 59
  Anti-HAV, ≤ 50 YOA | 4034.0 [2927.7 to 5558.4] | 1769.8 [1301.1 to 2407.3] | 5166.9 [3995.2 to 6682.2]
  Anti-HAV, 51-60 YOA: number analyzed (Participants) | 65 | 64 | 57
  Anti-HAV, 51-60 YOA | 2521.6 [1847.4 to 3441.7] | 1714.8 [1286.3 to 2286.0] | 3822.8 [2698.0 to 5416.4]
  Anti-HAV, ≥ 61 YOA: number analyzed (Participants) | 57 | 59 | 60
  Anti-HAV, ≥ 61 YOA | 2019.4 [1368.1 to 2980.9] | 873.8 [616.7 to 1237.9] | 2566.2 [1822.0 to 3614.4]
  Anti-HBs, ≤ 50 YOA: number analyzed (Participants) | 59 | 59 | 59
  Anti-HBs, ≤ 50 YOA | 1839.9 [1042.0 to 3248.9] | 753.7 [393.7 to 1443.1] | 217.2 [126.1 to 374.0]
  Anti-HBs, 51-60 YOA: number analyzed (Participants) | 65 | 64 | 57
  Anti-HBs, 51-60 YOA | 986.4 [583.1 to 1668.7] | 324.1 [182.6 to 575.3] | 286.6 [165.0 to 497.7]
  Anti-HBs, ≥ 61 YOA: number analyzed (Participants) | 57 | 59 | 60
  Anti-HBs, ≥ 61 YOA | 814.6 [425.2 to 1560.6] | 522.6 [262.7 to 1039.4] | 75.3 [40.9 to 138.6]

21. Secondary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations, by BMI
Description: Anti-HAV and anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL). The reference seropositivity cut-off values for anti-HAV and anti-HBs antibodies were equal to or above (≥) 15 mIU/mL and ≥ 3.3 mIU/mL, respectively. The antibody concentrations were stratified by BMI as follows: healthy, overweight and obese.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
mIU/mL
  Anti-HAV, Healthy: number analyzed (Participants) | 57 | 61 | 58
  Anti-HAV, Healthy | 3565.4 [2509.8 to 5065.1] | 1569.2 [1115.1 to 2208.4] | 4756.2 [3399.5 to 6654.5]
  Anti-HAV, Overweight: number analyzed (Participants) | 66 | 63 | 58
  Anti-HAV, Overweight | 2846.6 [2140.2 to 3786.3] | 1663.9 [1252.7 to 2210.1] | 3943.9 [2784.3 to 5586.4]
  Anti-HAV, Obese: number analyzed (Participants) | 58 | 58 | 60
  Anti-HAV, Obese | 1984.0 [1327.6 to 2964.9] | 1004.8 [718.8 to 1404.5] | 2716.2 [2065.6 to 3571.8]
  Anti-HBs, Healthy: number analyzed (Participants) | 57 | 61 | 58
  Anti-HBs, Healthy | 2140.5 [1168.9 to 3919.6] | 505.4 [274.1 to 931.8] | 475.2 [278.9 to 809.7]
  Anti-HBs, Overweight: number analyzed (Participants) | 66 | 63 | 58
  Anti-HBs, Overweight | 1540.8 [889.1 to 2670.2] | 609.4 [338.2 to 1097.9] | 165.9 [91.5 to 300.9]
  Anti-HBs, Obese: number analyzed (Participants) | 58 | 58 | 60
  Anti-HBs, Obese | 443.5 [268.5 to 732.7] | 368.3 [178.2 to 761.4] | 68.1 [41.9 to 110.7]

22. Secondary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations, by Smoking Status
Description: Anti-HAV and anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL). The reference seropositivity cut-off values for anti-HAV and anti-HBs antibodies were equal to or above (≥) 15 mIU/mL and ≥ 3.3 mIU/mL, respectively. The antibody concentrations were stratified by smoking status (smokers and non-smokers).
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
mIU/mL
  Anti-HAV, Smokers: number analyzed (Participants) | 51 | 51 | 32
  Anti-HAV, Smokers | 1844.6 [1233.7 to 2758.0] | 1433.2 [1012.9 to 2028.0] | 3456.0 [2363.5 to 5053.4]
  Anti-HAV, Non-Smokers: number analyzed (Participants) | 130 | 131 | 144
  Anti-HAV, Non-Smokers | 3216.5 [2578.8 to 4012.0] | 1379.2 [1106.8 to 1718.6] | 3766.3 [3047.8 to 4654.3]
  Anti-HBs, Smokers: number analyzed (Participants) | 51 | 51 | 32
  Anti-HBs, Smokers | 654.4 [358.8 to 1193.6] | 416.4 [204.4 to 848.2] | 108.1 [52.2 to 223.5]
  Anti-HBs, Non-smokers: number analyzed (Participants) | 130 | 131 | 144
  Anti-HBs, Non-smokers | 1438.3 [972.0 to 2128.5] | 525.5 [343.7 to 803.2] | 198.3 [136.6 to 288.0]

23. Secondary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations, by Alcohol Consumption
Description: Anti-HAV and anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL). The reference seropositivity cut-off values for anti-HAV and anti-HBs antibodies were equal to or above (≥) 15 mIU/mL and ≥ 3.3 mIU/mL, respectively. The antibody concentrations were stratified by alcohol consumption as follows: none or mild, moderate and heavy.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
mIU/mL
  Anti-HAV, None or Mild: number analyzed (Participants) | 112 | 106 | 102
  Anti-HAV, None or Mild | 2505.1 [1912.9 to 3280.7] | 1403.6 [1084.9 to 1816.0] | 3731.1 [2897.6 to 4804.2]
  Anti-HAV, Moderate: number analyzed (Participants) | 56 | 68 | 62
  Anti-HAV, Moderate | 3174.6 [2314.9 to 4353.6] | 1453.8 [1115.5 to 1894.7] | 3754.3 [2761.6 to 5103.8]
  Anti-HAV, Heavy: number analyzed (Participants) | 13 | 8 | 12
  Anti-HAV, Heavy | 3195.3 [1603.6 to 6366.8] | 899.8 [247.2 to 3274.9] | 3292.6 [1603.2 to 6762.1]
  Anti-HBs, None or Mild: number analyzed (Participants) | 112 | 106 | 102
  Anti-HBs, None or Mild | 1043.1 [689.5 to 1578.0] | 534.9 [339.9 to 841.7] | 230.7 [150.5 to 353.6]
  Anti-HBs, Moderate: number analyzed (Participants) | 56 | 68 | 62
  Anti-HBs, Moderate | 1136.7 [598.6 to 2158.5] | 467.3 [240.5 to 908.1] | 132.7 [72.6 to 242.4]
  Anti-HBs, Heavy: number analyzed (Participants) | 13 | 8 | 12
  Anti-HBs, Heavy | 3246.9 [1161.2 to 9078.8] | 223.4 [91.7 to 544.2] | 96.6 [27.3 to 341.8]

24. Secondary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations, by Concomitant Medication
Description: Anti-HAV and anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL). The reference seropositivity cut-off values for anti-HAV and anti-HBs antibodies were equal to or above (≥) 15 mIU/mL and ≥ 3.3 mIU/mL, respectively. The antibody concentrations were stratified by concomitant medication (concomitant medication and no concomitant medication).
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 165 | 169 | 162
mIU/mL
  Anti-HAV, concomitant medication | 2680.3 [2187.8 to 3283.7] | 1398.4 [1150.1 to 1700.2] | 3752.7 [3097.9 to 4546.0]
  Anti-HAV, no concomitant medication: number analyzed (Participants) | 16 | 13 | 14
  Anti-HAV, no concomitant medication | 3505.5 [1541.7 to 7971.1] | 1343.0 [801.0 to 2251.9] | 3225.1 [1470.3 to 7074.1]
  Anti-HBs, concomitant medication | 1138.0 [804.2 to 1610.3] | 533.4 [368.9 to 771.4] | 174.1 [124.6 to 243.3]
  Anti-HBs, no concomitant medication: number analyzed (Participants) | 16 | 13 | 14
  Anti-HBs, no concomitant medication | 1329.9 [405.9 to 4356.9] | 170.8 [30.3 to 962.4] | 255.8 [36.3 to 1803.6]

25. Secondary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations, by Medical Condition
Description: Anti-HAV and anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL). The reference seropositivity cut-off values for anti-HAV and anti-HBs antibodies were equal to or above (≥) 15 mIU/mL and ≥ 3.3 mIU/mL, respectively. The antibody concentrations were stratified by medical condition as follows: no medical condition, past medical condition and current medical condition.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 181 | 182 | 176
mIU/mL
  Anti-HAV,no medical condition: number analyzed (Participants) | 24 | 20 | 20
  Anti-HAV,no medical condition | 4765.5 [3301.7 to 6878.3] | 2187.5 [1387.0 to 3450.0] | 5531.9 [3806.7 to 8038.7]
  Anti-HAV,past medical condition: number analyzed (Participants) | 13 | 22 | 15
  Anti-HAV,past medical condition | 3438.3 [1944.8 to 6078.7] | 1882.2 [1275.1 to 2778.2] | 4073.9 [1915.1 to 8666.5]
  Anti-HAV,current medical condition: number analyzed (Participants) | 144 | 140 | 141
  Anti-HAV,current medical condition | 2445.3 [1935.9 to 3088.8] | 1245.2 [997.2 to 1554.8] | 3464.3 [2800.4 to 4285.7]
  Anti-HBs,no medical condition: number analyzed (Participants) | 24 | 20 | 20
  Anti-HBs,no medical condition | 2743.4 [1191.4 to 6316.9] | 435.2 [146.1 to 1296.7] | 345.1 [104.8 to 1136.5]
  Anti-HBs,past medical condition: number analyzed (Participants) | 13 | 22 | 15
  Anti-HBs,past medical condition | 1537.3 [316.0 to 7478.8] | 799.5 [292.4 to 2186.4] | 349.4 [117.6 to 1038.0]
  Anti-HBs,current medical condition: number analyzed (Participants) | 144 | 140 | 141
  Anti-HBs,current medical condition | 964.6 [668.1 to 1392.8] | 464.4 [304.0 to 709.5] | 152.2 [105.3 to 220.0]

26. Secondary Outcome: Number of Subjects With Anti-HAV and Anti-HBs Antibody Concentrations Above the Cut-off Value
Description: Seropositivity for anti-HAV antibodies was defined as anti-HAV antibody concentration equal to or above (≥) 15 mIU/mL and anti-HBs seropositivity was defined as anti-HBs antibody concentrations ≥ 3.3 mIU/mL. Anti-HBs AUSAB = anti-HBs antibody concentrations were tested with AUSAB EIA /Abbott assay; Anti-HBs in-house = anti-HBs antibody concentrations were tested with in-house assay (bridging).
Time Frame: At Month 12 (M12), Month 24 (M24) and Month 36 (M36)
Population: The analysis was performed Long Term According-To-Protocol (LT ATP) cohort for immunogenicity, which included all subjects who were included in the ATP cohort for immunogenicity in the primary study and who came within the blood sampling time interval at Months 12, 24 and 36.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 171 | 176 | 167
Participants
  Anti-HAV, M12: number analyzed (Participants) | 168 | 168 | 165
  Anti-HAV, M12 | 162 | 165 | 164
  Anti-HAV, M24: number analyzed (Participants) | 171 | 176 | 165
  Anti-HAV, M24 | 164 | 170 | 163
  Anti-HAV, M36: number analyzed (Participants) | 163 | 167 | 153
  Anti-HAV, M36 | 158 | 159 | 148
  Anti-HBs, M12 AUSAB: number analyzed (Participants) | 168 | 168 | 165
  Anti-HBs, M12 AUSAB | 153 | 134 | 109
  Anti-HBs, M24 AUSAB | 136 | 123 | 74
  Anti-HBs, M24 in-house: number analyzed (Participants) | 169 | 175 | 165
  Anti-HBs, M24 in-house | 137 | 129 | 76
  Anti-HBs, M36 in-house: number analyzed (Participants) | 163 | 167 | 153
  Anti-HBs, M36 in-house | 124 | 105 | 67

27. Secondary Outcome: Number of Seroprotected Subjects Against Hepatitis B Surface (HBs) Antigen
Description: A seroprotected subject was defined as a vaccinated subject with a serum anti-HBs antibody concentration equal to or above (≥) 10 mIU/mL. Anti-HBs AUSAB = anti-HBs antibody concentrations were tested with AUSAB EIA /Abbott assay; Anti-HBs in-house = anti-HBs antibody concentrations were tested with in-house assay (bridging).
Time Frame: At Month 12 (M12), Month 24 (M24) and Month 36 (M36)
Population: The analysis was performed on the LT ATP cohort for immunogenicity, which included all subjects who were included in the ATP cohort for immunogenicity in the primary study and who came within the blood sampling time interval at Months 12, 24 and 36.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 171 | 176 | 167
Participants
  Anti-HBs, M12 AUSAB: number analyzed (Participants) | 168 | 168 | 165
  Anti-HBs, M12 AUSAB | 147 | 124 | 93
  Anti-HBs, M24 AUSAB | 127 | 88 | 50
  Anti-HBs, M24 in-house: number analyzed (Participants) | 169 | 175 | 165
  Anti-HBs, M24 in-house | 125 | 99 | 56
  Anti-HBs, M36 in-house: number analyzed (Participants) | 163 | 167 | 153
  Anti-HBs, M36 in-house | 104 | 75 | 45

28. Secondary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations
Description: Anti-HAV and anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL). The reference seropositivity cut-off values for anti-HAV and anti-HBs antibodies were equal to or above (≥) 15 mIU/mL and ≥ 3.3 mIU/mL, respectively. Anti-HBs AUSAB = anti-HBs antibody concentrations were tested with AUSAB EIA /Abbott assay; Anti-HBs in-house = anti-HBs antibody concentrations were tested with in-house assay (bridging).
Time Frame: At Month 12 (M12), Month 24 (M24) and Month 36 (M36)
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 171 | 176 | 167
mIU/mL
  Anti-HAV, M12: number analyzed (Participants) | 168 | 168 | 165
  Anti-HAV, M12 | 891.0 [747.3 to 1062.2] | 530.6 [442.0 to 637.1] | 1200.5 [999.3 to 1442.1]
  Anti-HAV, M24 | 271.6 [229.0 to 322.2] | 209.9 [176.3 to 249.8] | 362.0 [303.5 to 431.8]
  Anti-HAV, M36: number analyzed (Participants) | 163 | 167 | 153
  Anti-HAV, M36 | 216.9 [182.6 to 257.6] | 185.4 [155.7 to 220.7] | 278.5 [229.4 to 338.2]
  Anti-HBs, M12 AUSAB: number analyzed (Participants) | 168 | 168 | 165
  Anti-HBs, M12 AUSAB | 339.2 [248.6 to 462.9] | 149.4 [106.4 to 209.7] | 53.1 [39.3 to 71.6]
  Anti-HBs, M24 AUSAB | 113.2 [83.9 to 152.8] | 46.5 [33.0 to 65.4] | 21.3 [15.5 to 29.4]
  Anti-HBs, M24 in-house: number analyzed (Participants) | 169 | 175 | 165
  Anti-HBs, M24 in-house | 99.3 [75.4 to 130.7] | 40.8 [30.4 to 54.9] | 22.3 [16.9 to 29.4]
  Anti-HBs, M36 in-house: number analyzed (Participants) | 163 | 167 | 153
  Anti-HBs, M36 in-house | 72.1 [53.1 to 98.0] | 34.1 [24.6 to 47.2] | 18.9 [14.1 to 25.3]

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Note: 3 subjects reported SAEs prior to administration of the first dose of vaccination.
Time Frame: From Day 0 up to Month 7
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 199 | 200 | 197
Participants | 11 | 14 | 16

30. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 29
Time Frame: At Month 12 (M12), Month 24 (M24) and Month 36 (M36)
Population: The analysis was performed on the Long Term Total Vaccinated Cohort, which included all subjects who had received at least one dose of the study vaccine in the primary study and who returned for the current blood sample time point at one, two and three years (Month 12, 24, 36) after first vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
Number analyzed (Participants) | 197 | 198 | 194
Participants
  Any SAE(s), M12 | 0 | 0 | 0
  Any SAE(s), M24: number analyzed (Participants) | 193 | 196 | 194
  Any SAE(s), M24 | 0 | 0 | 0
  Any SAE(s), M36: number analyzed (Participants) | 189 | 196 | 192
  Any SAE(s), M36 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs: from Day 0 up to Month 36.
Description: Only SAEs were collected during this study. Per Study Protocol, Other (non-serious) Adverse Events were not planned to be collected in this study.
Arm/Group | Twinrix Group | Engerix-B+Havrix Group | HB VAX PRO+Vaqta Group
All-Cause Mortality (participants affected / at risk) | 1/199 | 2/200 | 2/197
Serious Adverse Events (participants affected / at risk) | 11/199 | 14/200 | 16/197
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix Group (N=199) | Engerix-B+Havrix Group (N=200) | HB VAX PRO+Vaqta Group (N=197)
Pneumonia (Infections and infestations) | 0 | 0 | 2
Adams-Stokes syndrome (Cardiac disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Blepharochalasis (Eye disorders) | 0 | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastroduodenal ulcer (Blood and lymphatic system disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic neoplasm malignant (Hepatobiliary disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningitis (Infections and infestations) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 0
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Stress incontinence (Renal and urinary disorders) | 0 | 0 | 1
Subdural haematoma (Nervous system disorders) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.